CLINICAL TRIAL: NCT05461625
Title: Prospective, Randomized, Double Blinded Trial Comparing Clinical, Radiological and Laboratory Outcomes of Anterior Cruciate Ligament Reconstruction With or Without Concomitant AnteroLateral Ligament Reconstruction.
Brief Title: ACL Reconstruction With/Without ALL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, Professor CMKP, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACL_ALL
Record Dates: First submitted 2022-02-03; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: ACL Injury; ALL
Keywords: ACL, ALL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACL (Sham Comparator): Anterior cruciate ligament reconstruction without additional procedure
  Interventions: Procedure: ACL reconstruction
- ACL + ALL anatomic (Active Comparator): Anterior cruciate ligament reconstruction and anatomic anterolateral ligament reconstruction
  Interventions: Procedure: ACL reconstruction; Other: ALL anatomic
- ACL + ALL tenodesis (Active Comparator): Anterior cruciate ligament reconstruction and anterolateral ligament tenodesis
  Interventions: Procedure: ACL reconstruction; Other: ALL tenodesis

INTERVENTIONS:
Procedure: ACL reconstruction — Anterior cruciate ligament reconstruction
Other: ALL anatomic — anatomic anterolateral ligament reconstruction
  Arms: ACL + ALL anatomic
Other: ALL tenodesis — anterolateral ligament teondesis
  Arms: ACL + ALL tenodesis

SUMMARY:
This study will compare Anterior Cruciate Reconstruction with or without Anterolateral Ligament Reconstruction in patients with ACL injury. The purpose of this study is evaluate if addition of ALLr to ACLr provides better clinical, radiological and laboratory outcomes.

DETAILED DESCRIPTION:
This study compare ACL reconstruction and additional tenodesis or ALL recontruction described by Arnold. Patients will be randomized fot this tree group and surgeon will be blinded.

Anterolateral ligament reconstruction could play a role in augmenting rotational stability in the ACL-reconstructed knee and are most likely to benefit hyperlax patients, revision cases, pivoting athletes, and those with IKDC grade III pivot shifts. In our study we will would like to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

- primary ACL injury

Exclusion Criteria:

* no informed consent to participate in the study
* age under 18 years or above 65
* multilligament injury or single plane knee instability (medial, lateral)
* another musculoskeletal disorders in lower limb
* lower limb deformity requiring axis correction below 4o or above 12.5o
* joints inflammatory diseases
* ASA score > II

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 762 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Knee stability | 24 months
  KT-1000 assesment for knee stability

SECONDARY OUTCOMES:
Functional tests | 12 months
  hop-for-distance
KOOS (Knee injury and Osteoarthritis Outcome Score) | 6 weeks
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
KOOS (Knee injury and Osteoarthritis Outcome Score) | 6 months
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
KOOS (Knee injury and Osteoarthritis Outcome Score) | 24 months
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Tegner Lysholm Knee Scoring Scale | 6 weeks
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 6 months
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 24 months
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
IKDC (International Knee Documentation Committee) subjective knee evaluation | 6 weeks
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. highr number representing higher levels of function.
IKDC (International Knee Documentation Committee) subjective knee evaluation | 6 months
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. highr number representing higher levels of function.
IKDC (International Knee Documentation Committee) subjective knee evaluation | 24 months
  IKDC is subjective scale that provides patients with an overall function score. Total to a scaled number ranges from 0 to 100. highr number representing higher levels of function.
SF-36 (36-Item Short Form Survey) | 6 weeks
  Quality of life
SF-36 (36-Item Short Form Survey) | 6 months
  Quality of life
SF-36 (36-Item Short Form Survey) | 24 months
  Quality of life
VAS (Visual analog scale) | 6 weeks
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
VAS (Visual analog scale) | 6 months
  Pain Visual Analog Scale
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
VAS (Visual analog scale) | 24 months
  Pain Visual Analog Scale
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
KOOS PF (Knee injury and Osteoarthritis Outcome Score Patellofemoral) | 6 weeks
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability
KOOS PF (Knee injury and Osteoarthritis Outcome Score Patellofemoral) | 6 months
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability
KOOS PF (Knee injury and Osteoarthritis Outcome Score Patellofemoral) | 24 months
  the 'Knee Injury and Osteoarthritis Outcome Score Patellofemoral' questionnaire (KOOS-PF) is frequently used to measure symptoms and function among the people with PFJ-OA. This scale is scored from 0 to 100, with 100 representing no disability and 0 representing maximum disability

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Kaminski, Study Chair — SPSK CMKP
Locations (1):
- Department of Orthopaedics and Traumatology, Centre of Postgraduate Medical Education, Professor A. Gruca Teaching Hospital, Otwock, Masovian Voivodeship, Poland